CLINICAL TRIAL: NCT06069778
Title: A Phase I/Randomized Phase II, Open-label Multicenter Trial to Evaluate the Safety, Tolerability, and Efficacy of mFOLFIRINOX With or Without BNT321 as Adjuvant Therapy Following Curative Resection in Patients With Pancreatic Adenocarcinoma
Brief Title: Safety, Tolerability, and Efficacy of mFOLFIRINOX ± BNT321 as Adjuvant Therapy Following Curative Resection in Patients With Pancreatic Adenocarcinoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: BioNTech SE (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: BNT321-02; 2023-506014-47 (EudraCT Number)
Record Dates: First submitted 2023-09-11; First posted 2023-10-06 (Actual); Results first posted 2025-10-31 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Pancreatic Cancer
Keywords: CA19-9 Positive Malignancies; Pancreatic Cancer and other CA19-9 expressing malignancies; Pancreatic Ductal Adenocarcinoma (PDAC); Sialyl Lewis A (sLea)
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Radiologists that assess the CT scans will be blinded to the study treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase 1 - BNT321 0.5 mg/kg + mFOLFIRINOX (Experimental): BNT321 in combination with mFOLFIRINOX chemotherapy (24 weeks) followed by BNT321 monotherapy (24 weeks)
  Interventions: Drug: BNT321 0.5 mg/kg; Drug: mFOLFIRINOX
- Phase 1 - BNT321 DL 2 + mFOLFIRINOX (Experimental): BNT321 in combination with mFOLFIRINOX chemotherapy (24 weeks) followed by BNT321 monotherapy (24 weeks)
  Interventions: Drug: BNT321 DL 2; Drug: mFOLFIRINOX
- Phase 2 - BNT321 RP2D + mFOLFIRINOX (Experimental): BNT321 in combination with mFOLFIRINOX chemotherapy (24 weeks) followed by BNT321 monotherapy (24 weeks)
  Interventions: Drug: mFOLFIRINOX; Drug: BNT321 RP2D
- Phase 2 - mFOLFIRINOX (Active Comparator): mFOLFIRINOX chemotherapy (24 weeks) as monotherapy
  Interventions: Drug: mFOLFIRINOX

INTERVENTIONS:
Drug: BNT321 0.5 mg/kg — Intravenous infusion
  Arms: Phase 1 - BNT321 0.5 mg/kg + mFOLFIRINOX
Drug: BNT321 DL 2 — Intravenous infusion
  Arms: Phase 1 - BNT321 DL 2 + mFOLFIRINOX
Drug: mFOLFIRINOX — Intravenous infusion
Drug: BNT321 RP2D — Intravenous infusion
  Arms: Phase 2 - BNT321 RP2D + mFOLFIRINOX

SUMMARY:
This study was designed as a Phase 1/randomized Phase 2 open-label study of modified(m) FOLFIRINOX ± BNT321 for adjuvant therapy in pancreatic ductal adenocarcinoma (PDAC) patients post R0 or R1 resection.

The Phase 1, dose escalation part of this study was planned to be a limited evaluation of two planned BNT321 dose levels (DLs) in combination with mFOLFIRINOX chemotherapy (24 weeks) followed by BNT321 monotherapy (24 weeks). Following completion of the dose escalation Phase 1 and identification of the recommended Phase 2 dose (RP2D), the study was designed as a 2-arm, randomized Phase 2 of mFOLFIRINOX ± BNT321 to evaluate the efficacy of mFOLFIRINOX + BNT321 versus mFOLFIRINOX alone as adjuvant therapy in PDAC patients post R0 or R1 resection. Treatment cycles were every 2 weeks (14 days).

DETAILED DESCRIPTION:
The Phase 1 part of the study was planned to be a limited dose finding evaluation, whereby a minimal number of BNT321 DLs were planned to be tested for safety and tolerability in combination with mFOLFIRINOX chemotherapy. Dose escalation was planned to be conducted using a 3+3 design, with up to six additional participants treated at the Phase 1 defined combination maximum tolerated dose (MTD). Two BNT321 DLs were initially planned, 0.5 mg/kg and a second DL 2. Following evaluation of safety profile for DL 2, additional BNT321 DLs could have been evaluated following safety data review, discussion, and approval by the safety review committee (SRC), and health authority review and approval. Approximately 20 participants were planned to be enrolled into the Phase 1 part.

Following completion of the dose escalation Phase 1 and identification of the RP2D, the study was planned to proceed to a randomized Phase 2 part. For this part, an independent data monitoring committee was planned to be be established prior to the inclusion of the first participant in this phase.

The randomized Phase 2 was designed to enroll up to 300 participants to enable a robust statistical evaluation of the study's Phase 2 primary endpoint, i.e., median disease-free survival (mDFS).

Additional evaluations for Phase 2 were planned to include determination of combination regimen safety and tolerability, determination of overall survival (OS), pharmacokinetic (PK), and pharmacodynamic (PD) analyses including anti-drug antibody (ADA), complement-dependent cytotoxicity (CDC), antibody-dependent cell-mediated cytotoxicity (ADCC) assessments, cytokine and circulating tumor DNA (ctDNA) assessments.

The study was terminated early by the sponsor due to strategic reprioritization and not due to safety concerns. At the time of the termination, only one dose level (i.e., 0.5 mg/kg) of BNT321 was tested.

ELIGIBILITY:
Inclusion Criteria:

* Has signed an informed consent form (ICF) before initiation of any study-specific procedures
* Was >18 years or age deemed to be an adult per local authorities inclusive, at the time of giving written informed consent
* Were willing and able to comply with scheduled visits, treatment schedule, laboratory tests, lifestyle restrictions, and other requirements of the study (per investigator assessment, must been capable of understanding and following study-related instructions)
* Had an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1
* Had histologically or cytologically confirmed PDAC
* Had macroscopically complete resection (R0 or R1 resection, Royal College of Pathologists [RCP] classification) performed between ≥21 and ≤84 days prior to Cycle 1, Day 1 (C1D1). Submission of formalin-fixed paraffin-embedded tissue (FFPE) tumor tissue from resection or biopsy was required
* Had no radiologic (computed tomography/magnetic resonance imaging) evidence of metastatic disease, malignant ascites, or pleural effusion through an assessment obtained within 4 weeks of first study medication (i.e., C1D1)
* Full recovery from surgery and able to receive chemotherapy
* Had acceptable laboratory parameters
* Was willing to allow collection of pharmacokinetic samples
* Agreed not to enroll in another study of an IMP, starting after signing of the ICF and continuously until the last planned visit in this study
* Participants of childbearing potential (POCBP) must not been pregnant. POCBP, male participants who were sexually active with POCBP, and female partners of male participants should have used a highly effective method of contraception continuously throughout the study and for a period of 111 days after the last dose of BNT321 and for 9 months (POCBP) and 6 months (male participants) after the last oxaliplatin dose
* POCB who agreed not to donate eggs (ova, oocytes) starting after signing of the ICF and continuously throughout the study and for a period of 3 months after the last dose of BNT321 and for 9 months after the last oxaliplatin dose
* Men who were willing to refrain from sperm donation, starting after signing of ICF and continuously throughout the study until 111 days after receiving the last dose of BNT321 and for 6 months after the last oxaliplatin dose

Exclusion Criteria:

* Participants were pregnant or breastfeeding or planning pregnancy or to father children during the study or within 60 days after last IMP treatment
* A medical, psychological, or social condition which, in the opinion of the investigator, could have compromised their wellbeing if they participated in the study, or that could have prevented, limited, or confounded the protocol specified assessments or procedures, or that could have impacted adherence to protocol-described requirements
* Had major surgery within 3 weeks of first dose of the study treatment, where participation in the study could have compromised the participant's wellbeing in the opinion of the investigator
* Had abnormal electrocardiograms (ECGs) that were clinically significant, such as Fridericia-corrected QT prolongation >470 msec (for women) and >450 msec (for men), (average of three ECGs at least 5 minutes apart)
* Had a history of anaphylactic reaction to human, or humanized, antibody
* Have had other known active cancer(s) likely to require treatment in the next 2 years
* Had prior radiotherapy or systemic treatment for PDAC
* Active, uncontrolled bacterial, viral, or fungal infection(s) requiring systemic antiinfective therapy that has been administered less than 2 weeks prior to the first dose of BNT321
* Known hypersensitivity to any of the excipients of the experimental product BNT321
* Known history of seropositivity for human immunodeficiency virus (HIV) with CD4+ T-cell counts <350 cells/μL and with a history of acquired immunodeficiency syndrome (AIDS)-defining opportunistic infections
* Known history/positive serology for Hepatitis B requiring active antiviral therapy (unless immune due to vaccination or resolved natural infection or unless passive immunization due to immunoglobulin therapy; participants with positive serology must have had Hepatitis B virus viral load below the limit of quantification)
* Active Hepatitis C virus infection (participants who have had completed curative antiviral treatment with Hepatitis C virus viral load below the limit of quantification were allowed)
* Use of any IMP or device within 21 days before administration of first dose of study treatment or ongoing participation in the active treatment phase of another interventional clinical study
* Was subject to exclusion periods from another investigational study
* Were vulnerable individuals as per ICH E6 definition, i.e., individuals whose willingness to participate in a clinical study may be unduly influenced by the expectation, whether justified or not, of benefits associated with participation, or of a retaliatory response from senior members of a hierarchy in case of refusal to participate.
* Serum CA19-9 >180 U/mL within 3 weeks of C1D1
* Incomplete macroscopic tumor removal (R2 resection)
* Significant cardiovascular risk (past medical history of coronary stenting or myocardial infarction within 6 months, or New York Heart Association (NYHA) Class III/IV, heart failure, or concurrent unstable angina) or risk factors for QT prolongation (sustained Grade 3 or higher hypokalemia, history of unstable arrhythmia or family history of long QT syndrome)
* Pre-existing neuropathy
* Homozygous UDP glucuronosyltransferase family 1 member A1 (UGT1A1)*28 mutation, if testing was required by local regulations
* Inflammatory disease of the colon or rectum, or occlusion or sub-occlusion of the intestine or severe post-operative uncontrolled diarrhea
* Complete dihydropyrimidine dehydrogenase deficiency, if testing was required by local regulations
* Received a live vaccine within 3 weeks prior to the first dose of study treatment
* Participants with a contraindication to receiving mFOLFIRINOX
* Participants with active or latent tuberculosis or history of Mycobacterium tuberculosis infection currently or within the last 2 years
* Individuals committed to an institution by virtue of an order issued either by the judicial or the administrative authorities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2024-03-27 (Actual); Primary Completion 2024-09-18 (Actual); Study Completion 2024-09-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: BioNTech Responsible Person, Study Director — BioNTech SE
Locations (2):
- United States (2):
  - Valkyrie Clinical Trials, Los Angeles, California
  - Medical University of South Carolina (MUSC), Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1 - BNT321 0.5 mg/kg + mFOLFIRINOX: BNT321 in combination with mFOLFIRINOX chemotherapy. mFOLFIRINOX: Administered as intravenous infusion on the first day of each 14-day cycle (i.e., C1D1, C2D1, C3D1, and so on for a total of 12 cycles) using the following agent, oxaliplatin (Day 1), leucovorin (Day 1), irinotecan (Day 1, starting 30 minutes after leucovorin), and 5-fluorouracil (Day 1).
  BNT321: Administered as intravenous infusion and incorporated into the mFOLFIRINOX regimen starting from the second cycle and after the completion of the 5-fluorouracil infusion (e.g., initially on C2D3).
Period: Overall Study
Arm/Group | Phase 1 - BNT321 0.5 mg/kg + mFOLFIRINOX
Started | 1
Completed | 0
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Analysis was performed on the safety set that included all participants who received at least one dose of the investigational medicinal product (IMP).
Arm/Group | Phase 1 - BNT321 0.5 mg/kg + mFOLFIRINOX
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 1
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Not disclosed to avoid re-identification | 1
Race/Ethnicity, Customized [Number; unit: participants]
  Not disclosed to avoid re-identification | 1
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Phase 1 - The Number and Percentage of Participants With at Least One Dose of Investigational Medicinal Product (IMP) Reporting Treatment Emergent Adverse Events (TEAEs)
Description: TEAEs graded per Common Toxicity Criteria for Adverse Events version 5.0 (CTCAE v5.0), including Grade ≥3, serious, fatal TEAE by relationship.
Time Frame: from the start of study drug treatment until the end of study (i.e., 164 days)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 - BNT321 0.5 mg/kg + mFOLFIRINOX
Number analyzed (Participants) | 1
Participants | 1

2. Primary Outcome: Phase 1 - The Number and Percentage of Participants With at Least One Dose of IMP Reporting Occurrence of Dose Limiting Toxicities (DLTs)
Description: For all Phase I cohorts the DLT assessment period was planned to encompass the treatment cycles of the first two consecutive BNT321 doses, i.e., 28 days within treatment Cycles 2 and 3.
  To be considered a DLT, an AE must have met the following three criteria:
  * Occurred during the DLT assessment period of BNT321.
  * Was considered BNT321-related (i.e., definitely related or possibly related).
  * Occurred in the presence of adequate supportive care (e.g., Grade 3 vomiting despite use of an appropriate anti-emetic regimen).
  In addition, to be considered a DLT, an AE must have met at least one of the additional criteria using CTCAE v5.0 as specified in the protocol.
Time Frame: up to 28 days after first dose of BNT321
Population: The participant was not evaluable for DLT due to not satisfying the minimum exposure criterion as defined in the protocol.
Arm/Group | Phase 1 - BNT321 0.5 mg/kg + mFOLFIRINOX
Number analyzed (Participants) | 0

3. Primary Outcome: Phase 2 - Disease-free Survival (DFS)
Description: DFS was defined as the time from randomization to occurrence of any of the following events, whichever occurs first:
  * Locoregional recurrence or distant metastases as determined by an independent central radiology assessment.
  * Occurrence of second primary (same or other) cancer as determined by an independent central radiology assessment.
  * Death from any cause.
Time Frame: up to 60 months
Population: Due to early termination of the study, no participant was included in the Phase 2 part of the study.
Arm/Group | Phase 2 - BNT321 RP2D + mFOLFIRINOX | Phase 2 - mFOLFIRINOX
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Phase 1 and 2 - OS
Description: OS was defined as the time from first dose of study treatment to death from any cause.
Time Frame: up to 60 months
Population: Data were not available for this endpoint, due to early termination of the study after enrollment of one participant in the Phase 1 part. The participant was followed up for efficacy for a short period of time while on study (~6 months), therefore there was insufficient data for the Phase 1 part to conduct a meaningful assessment of OS.
  No participant was included in the Phase 2 part of the study.
Arm/Group | Phase 1 - BNT321 0.5 mg/kg + mFOLFIRINOX
Number analyzed (Participants) | 0

5. Secondary Outcome: Phase 1 and 2 - Relapsed Free Survival (RFS)
Description: RFS is defined as the time from randomization to occurrence of any of the following events, whichever occurs first:
  * Locoregional recurrence or distant metastasis as determined by the investigator.
  * Death from any cause.
Time Frame: up to 60 months
Population: Data were not available for this endpoint, due to early termination of the study after enrollment of one participant in the Phase 1 part. The participant was followed up for efficacy for a short period of time while on study (~6 months) and disease was not relapsed, therefore there was insufficient data for the Phase 1 part to conduct a meaningful assessment of RFS.
  No participant was included in the Phase 2 part of the study.
Arm/Group | Phase 1 - BNT321 0.5 mg/kg + mFOLFIRINOX
Number analyzed (Participants) | 0

6. Secondary Outcome: Phase 1 and 2 - PK Assessments: Mean Area Under the Curve (AUC) Values Derived From Serum Concentration of IMP
Description: Mean AUC from participants who are dosed with at least one dose of IMP and who have evaluable PK data in Cycles 2 and 3 followed by sparse sampling through end of study (EOT).
Time Frame: up to 48 weeks
Population: Data were not available for this endpoint, due to early termination of the study after enrollment of one participant in the Phase 1 part. Therefore there was insufficient data for the Phase 1 part to conduct a meaningful assessment of the mean AUC.
  No participant was included in the Phase 2 part of the study.
Arm/Group | Phase 1 - BNT321 0.5 mg/kg + mFOLFIRINOX
Number analyzed (Participants) | 0

7. Secondary Outcome: Phase 1 and 2 - PK Assessments: Mean Observed Maximum Concentration (Cmax) Derived From Serum Concentration of IMP
Description: Mean Cmax from participants who are dosed with at least one dose of IMP and who have evaluable PK data in Cycles 2 and 3 followed by sparse sampling through EOT.
Time Frame: up to 48 weeks
Population: Data were not available for this endpoint, due to early termination of the study after enrollment of one participant in the Phase 1 part. Therefore there was insufficient data for the Phase 1 part to conduct a meaningful assessment of Cmax.
  No participant was included in the Phase 2 part of the study.
Arm/Group | Phase 1 - BNT321 0.5 mg/kg + mFOLFIRINOX
Number analyzed (Participants) | 0

8. Secondary Outcome: Phase 1 and 2 - PK Assessments: Median Time to Reach Cmax (Tmax) Derived From Serum Concentration of IMP
Description: Median tmax from participants who are dosed with at least one dose of IMP and who have evaluable PK data in Cycles 2 and 3 followed by sparse sampling through EOT.
Time Frame: up to 48 weeks
Population: Data were not available for this endpoint, due to early termination of the study after enrollment of one participant in the Phase 1 part. Therefore there was insufficient data for the Phase 1 part to conduct a meaningful assessment of Tmax.
  No participant was included in the Phase 2 part of the study.
Arm/Group | Phase 1 - BNT321 0.5 mg/kg + mFOLFIRINOX
Number analyzed (Participants) | 0

9. Secondary Outcome: Phase 1 and 2 - Percentage of Participants With Detectable Anti-drug Antibody (ADA)
Description: Percentage of participants who are dosed with at least one dose of IMP and with detectable ADA formation in Cycles 1 and 3, followed by sparse sampling through EOT
Time Frame: up to 48 weeks
Population: Data were not available for this endpoint, due to early termination of the study after enrollment of one participant in the Phase 1 part. The participant was followed up for a short period of time while on study (~6 months), therefore there was insufficient data for the Phase 1 part to conduct a meaningful assessment of detectable ADA.
  No participant was included in the Phase 2 part of the study.
Arm/Group | Phase 1 - BNT321 0.5 mg/kg + mFOLFIRINOX
Number analyzed (Participants) | 0

10. Secondary Outcome: Phase 1 and 2 - Percentage of Participants With Detectable and Durable ADCC and/or CDC Activity
Description: Percentage of participants who are dosed with at least one dose of IMP with detectable and durable (measurable throughout time on study) ADCC and/or CDC activity in Cycles 2 and 4, followed by sparse sampling through EOT
Time Frame: up to 48 weeks
Population: Data were not available for this endpoint, due to early termination of the study after enrollment of one participant in the Phase 1 part. The participant was followed up for a short period of time while on study (~6 months), therefore there was insufficient data for the Phase 1 part to conduct a meaningful assessment of detectable and durable ADCC and/or CDC activity No participant was included in the Phase 2 part of the study.
Arm/Group | Phase 1 - BNT321 0.5 mg/kg + mFOLFIRINOX
Number analyzed (Participants) | 0

11. Secondary Outcome: Phase 1 and 2 - Change From Baseline for Participant-reported Health-related Quality of Life (HRQoL) Using the European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Core Questionnaire (QLQ-C30)
Description: Change from baseline at end of Cycle 12 for participant-reported HRQoL using EORTC QLQ-C30
Time Frame: up to 60 months
Population: Data were not available for this endpoint, due to early termination of the study after enrollment of one participant in the Phase 1 part. The participant was followed up for efficacy for a short period of time while on study (~6 months), therefore there was insufficient data for the Phase 1 part to conduct a meaningful assessment of HRQoL.
  No participant was included in the Phase 2 part of the study.
Arm/Group | Phase 1 - BNT321 0.5 mg/kg + mFOLFIRINOX
Number analyzed (Participants) | 0

12. Secondary Outcome: Phase 1 and 2 - Change From Baseline for Participant-reported HRQoL Using EORTC Quality of Life Questionnaire for Pancreatic Cancer (QLQ-Pan26) Questionnaires
Description: Change from baseline at end of Cycle 12 for participant-reported HRQoL using EORTC QLQ-Pan26 questionnaires
Time Frame: up to 60 months
Population: as for outcome 11
Arm/Group | Phase 1 - BNT321 0.5 mg/kg + mFOLFIRINOX
Number analyzed (Participants) | 0

13. Secondary Outcome: Phase 1 and 2 - Change From Baseline in Combined Item Scores From EORTC QLQ-C30
Description: Change from baseline at end of Cycle 12 in combined item scores from EORTC QLQ-C30
Time Frame: up to 60 months
Population: as for outcome 11
Arm/Group | Phase 1 - BNT321 0.5 mg/kg + mFOLFIRINOX
Number analyzed (Participants) | 0

14. Secondary Outcome: Phase 1 and 2 - Change From Baseline in Combined Item Scores From EORTC QLQ-Pan26
Description: Change from baseline at end of Cycle 12 in combined item scores from EORTC QLQ-Pan26.
Time Frame: up to 60 months
Population: as for outcome 11
Arm/Group | Phase 1 - BNT321 0.5 mg/kg + mFOLFIRINOX
Number analyzed (Participants) | 0

15. Secondary Outcome: Phase 2 - Occurrence of TEAEs Including Grade ≥3, Serious, Fatal TEAE by Relationship
Time Frame: up to 12 months
Population: Due to early termination of the study, no participant was included in the Phase 2 part of the study.
Arm/Group | Phase 2 - BNT321 RP2D + mFOLFIRINOX | Phase 2 - mFOLFIRINOX
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Phase 2 - Occurrence of Dose Reduction and Discontinuation of IMP Due to TEAE
Description: Occurrence within a participant.
Time Frame: up to 12 months
Population: Due to early termination of the study, no participant was included in the Phase 2 part of the study.
Arm/Group | Phase 2 - BNT321 RP2D + mFOLFIRINOX | Phase 2 - mFOLFIRINOX
Number analyzed (Participants) | 0 | 0

17. Secondary Outcome: Phase 2 - Occurrence of Abnormal Laboratory Parameters
Description: Occurrence within a participant.
Time Frame: up to 48 weeks
Population: Due to early termination of the study, no participant was included in the Phase 2 part of the study.
Arm/Group | Phase 2 - BNT321 RP2D + mFOLFIRINOX | Phase 2 - mFOLFIRINOX
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Deaths and serious adverse events (SAEs): All events from the signing of the study-specific informed consent from until the end of study (i.e., 175 days). Other adverse events (AEs): All TEAEs, i.e., AEs reported from the start of study drug treatment until the end of study (i.e., 164 days).
Description: Other AEs: All TEAEs, i.e., AEs with an onset date on or after the first dose of the IMP (if the AE was absent before the first dose) or worsened after the first dose of IMP (if the AE was present before the first dose). AEs with an onset date >60 days after the last dose of IMP are included only if assessed as related to the IMP by the investigator.
Arm/Group | Phase 1 - BNT321 0.5 mg/kg + mFOLFIRINOX
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1 - BNT321 0.5 mg/kg + mFOLFIRINOX (N=1)
Alanine aminotransferase increased (Investigations) | 1
Blood alkaline phosphatase increased (Investigations) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Aspartate aminotransferase increased (Investigations) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Conjunctivitis (Infections and infestations) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hyperphosphataemia (Metabolism and nutrition disorders) | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1
Lymphocyte count decreased (Investigations) | 1
Lymphocyte count increased (Investigations) | 1
Nausea (Gastrointestinal disorders) | 1
Neutrophil count decreased (Investigations) | 1
Neuropathy peripheral (Nervous system disorders) | 1
Pharyngitis (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigators respectively trial sites shall not publish or refer to in writing or orally, in whole or in part, any data, information or materials generated from the study and the services, without the prior written consent of the sponsor.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-22): https://cdn.clinicaltrials.gov/large-docs/78/NCT06069778/Prot_SAP_000.pdf